CLINICAL TRIAL: NCT02994888
Title: PROSPECT-C: A Prospective Translational Study Investigating Molecular Predictors of Resistance and Response to Cetuximab or Panitumumab in Metastatic Colorectal Cancer
Brief Title: PROSPECT-C: A Study of Biomarkers of Response or Resistance to Anti-EGFR Therapies in Metastatic Colorectal Cancer
Acronym: PROSPECT-C
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3770
Record Dates: First submitted 2013-05-30; First posted 2016-12-16 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Both fresh frozen tissue and formalin-fixed paraffin-embedded (FFPE) tissue samples will be obtained. In addition, the following blood samples will also be taken;
  1. Baseline: an initial 20mL research blood sample (EDTA or equivalent (CPT) tube) will be collected
  2. Every 4 weeks until disease progression or patient death: 1 x 10mL research blood sample (EDTA or equivalent (CPT) tube) will be collected
  3. At time of progressive disease: final 10mL research blood sample (EDTA or equivalent (CPT) tube)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all patients: All patients will be treated with cetuximab 500mg/m2 every 2 weeks until the time of progression
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — All patients will be offered cetuximab 500mg/m2 every 2 weeks, until the time of progression

SUMMARY:
PROSPECT-C is a phase II study investigating the molecular markers of response or resistance to anti-epidermal growth factor receptor (EGFR) antibodies.

DETAILED DESCRIPTION:
Cetuximab or panitumumab are two monoclonal antibodies that are routinely offered to patients with metastatic colorectal cancer when they have no mutation in RAS genes. In Royal Marsden Hospital patients, who are refractory to all standard therapies and have metastatic colorectal cancer are offered one of these agents in third line metastatic setting. Whilst the mechanisms of response/resistance to these therapies are well studies, they are still incompletely understood. The main hypothesis of this study is that finding mechanisms of response and/or resistance by using novel techniques such as next generation sequencing (NGS) and/or digital droplet polymerase chain reaction (ddPCR) to these therapies will allow better patient selection and application of precision medicine in such patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients with a histologically confirmed diagnosis of metastatic colorectal adenocarcinoma
2. wild-type RAS tumour status by molecular analysis at the Royal Marsden Hospital
3. patients with inoperable metastatic colorectal cancer who are scheduled to be treated with cetuximab (or panitumumab) either as monotherapy or in combination with chemotherapy with palliative intent
4. patients who have received prior treatment with oxaliplatin, irinotecan and fluoropyrimidine containing chemotherapy regimens OR intolerance/contraindication to either oxaliplatin or irinotecan based chemotherapy, and planned to receive retreatment with EGFR monoclonal antibody (mAB) monotherapy or with EGFR mAB combined with a chemotherapy (irinotecan or oxaliplatin-based) that a patient has already received for a minimum of 3 months during a previous line of therapy.
5. patients who have metastatic disease sites which are amenable to core biopsy (preferably liver, soft tissue or nodal disease, with at least one lesion 3cm or more in diameter. If largest lesion 2-3cm diameter, eligibility to be discussed with radiologist prior to study entry)
6. patients aged 18 years or older
7. able to provide fully informed consent, to comply with the trial and follow-up procedures
8. receiving treatment at the Royal Marsden Hospital

Exclusion Criteria:

1. patients who have previously received treatment with cetuximab or panitumumab
2. previous malignancy other than colorectal cancer in the past 5 years, other than pre-invasive malignancy of the cervix or basal cell carcinoma, EXCEPT when the patient has histological confirmation of metastatic colorectal cancer at the site that is planned to be biopsied at baseline and on progression of disease
3. patients who are being anti-coagulated with warfarin or heparin
4. Patients that are participating in another clinical trial involving an investigational medicinal product, unless it is more than 14 days after they have ceased the investigational medicinal product
5. Patients that are participating in another research study involving tumour tissue biopsies planned to take place during the time that the patient is participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a histologically confirmed diagnosis of metastatic colorectal adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2012-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Track and validate specific known mechanisms of resistance/response to anti-EGFR therapies through | 3-4 years
  digital droplet polymerase chain reaction (ddPCR) and ultra deep next generation sequencing (NGS) analyses of circulating tumour deoxyribonucleic acid (ct-DNA) obtained every 4 weeks during the course of treatment. Mutations found in ctDNA will also be analysed in the archival and fresh tissue specimens, used for diagnostic testing and obtained during the study respectively

SECONDARY OUTCOMES:
Identify novel biomarkers of resistance to anti-EGFR therapies through whole exome sequencing | 3-4 years
  DNA extracted from pre- and post-treatment metastatic colorectal cancer (mCRC) biopsies; Ultra deep targeted sequencing of tumour samples and of ctDNA will be used to assess whether the identified resistance biomarkers are detectable in some patients before treatment initiation and whether this correlates with short progression free survival (PFS) and poor radiological response

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Surrey, Sutton, United Kingdom